CLINICAL TRIAL: NCT05465616
Title: Efficacy of Viome's Precision Nutrition Program Towards Reducing HbA1c
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V197
Record Dates: First submitted 2022-07-08; First posted 2022-07-20 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Diabetes; Pre Diabetes
Keywords: Health; Wellness; Nutrition; Vitamins; Supplements; Prebiotics; Probiotics; Fitness; Blood sugar
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded for this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (No Intervention): Participants with HbA1c levels between 5.7-8.9% (inclusive) are randomized into this arm. They may be provided with any combination of nutritional recommendations and supplements. Placebo capsules will contain inert and inactive materials. Participants may need to use a mobile app in order to participate in the trial.
- Viome's Precision Nutrition Program (VPNP) (Experimental): Participants with HbA1c levels between 5.7-8.9% (inclusive) are randomized into this arm. They may be provided with any combination of nutritional recommendations and supplements. Participants may need to use a mobile app in order to participate in the trial.
  Interventions: Dietary Supplement: Viome's Precision Nutrition Program (VPNP)

INTERVENTIONS:
Dietary Supplement: Viome's Precision Nutrition Program (VPNP) — Nutrition, diet, and possible coaching through Viome application. Precision supplement based on the participants microbiome sample results.
  Arms: Viome's Precision Nutrition Program (VPNP)

SUMMARY:
This is a randomized, placebo-controlled trial that will test the efficacy of VPNP in reducing HbA1c. Participant recruitment will occur through direct-to-participant enrollment. No additional clinical sites will be used for recruitment.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled trial that will test the efficacy of VPNP in reducing HbA1c. Participants with HbA1c levels between 5.7-8.9% (inclusive) will be recruited and randomized into either the placebo or intervention group. The study duration for each participant will be approximately 90 days. At the beginning of the 90 days, the participant will complete online questionnaires, a blood draw, and a set of at-home sample collections for blood, stool, and saliva that will be sent back to Viome. After the samples are analyzed, the participant will receive dietary recommendations (either personalized or USDA) and supplements (either personalized or placebo). The participant will follow the dietary recommendations and take the supplements for 90 days. At the end of the 90 days, the participant will once again complete online questionnaires, a blood draw, and a set of at-home sample collections for blood, stool, and saliva that will be sent back to Viome for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form and medical release prior to any trial-specific procedures are performed
* Females and males aged 18 years or older
* Able to speak and read English
* HbA1c between 5.7-8.9% (inclusive), tested within the past 30 days
* Willing and able to visit a Quest Diagnostic Patient Service Center (PSC)
* Willing and able to follow the trial instructions and Viome's Precision Nutrition Program
* Willing and able to use a smartphone and Viome app.

Exclusion Criteria:

* Antibiotic use within one month of the GI test
* Gestation within previous 6 month
* Current (or previous) use of medications that increase insulin (sulfonylureas, such as glimepiride, glipizide, glyburide, etc.)
* Current (or previous) use of exogenous insulin (such as Tresiba, Lantus, Toujeo, Levemir, Humalog, Novolog, Apidra, Fiasp, etc.)
* On a specific diet, such as ketogenic, for the purpose of reducing HbA1c and/or weight within the previous month
* Taking diet pills
* Allergy to an ingredient in the MH capsule or stick pack
* Currently on an investigational product
* Significant surgery or medical procedure planned
* Diet or lifestyle change during the trial period, besides those appropriate for trial arm Has followed Viome nutritional recommendations (foods and/or supplements)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-12-13 (Estimated); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
HbA1c Levels | 4 months
  HbA1c changes in individuals in the interventional arm compared to baseline measurement.
Insulin Resistance | 4 months
  Change in fasting insulin levels in those in the interventional arm compared to baseline measurement.

SECONDARY OUTCOMES:
BMI | 4 months
  Changes in BMI of individuals in the interventional arm compared to baseline measurement.
Cholesterol | 4 months
  Changes in HDL, LDL, total cholesterol, and triglyceride levels of those in the interventional arm compared to baseline measurements.
Waist to Hip Ratio | 4 months
  Changes in waist to hip ratio of those in the interventional group compared to baseline measurement.
Cardiovascular Risk | 4 months
  Changes to 10 year cardiovascular risk score of those in the interventional arm compared to baseline score.
Patient Health Questionnaire 9 (PHQ 9) Score | 4 months
  Changes in PHQ9 score of those in the interventional arm compared to baseline answers. The minimum PHQ 9 score is 0 and the maximum PHQ 9 score is 27. Higher scores indicate a worse outcome.
General Anxiety Disorder - 7 Score | 4 months
  Changes in GAD7 score in those in the interventional arm compared to baseline assessment. The minimum score on GAD 7 is 0-4 indicating none to minimal anxiety and the maximum score is 15-21 indicating sever anxiety. Higher scores indicate a worse outcome.
Species prevalence in stool, blood, and saliva | 4 months
  Changes in the prevalence of species in stool, blood, and saliva samples compared to baseline analysis.
Fasting glucose | 4 months
  Fasting glucose changes in individuals in the interventional arm compared to baseline measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, Principal Investigator — Viome
Locations (1):
- Viome Life Sciences, Bothell, Washington, United States